CLINICAL TRIAL: NCT00943046
Title: Master Study of the SIELLO Pacemaker Leads
Brief Title: Master Study for the Investigation of Safety and Efficacy of the SIELLO Pacemaker Leads
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 43-1
Record Dates: First submitted 2009-07-14; First posted 2009-07-21 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2017-05

CONDITIONS: Cardiac Pacemaker Syndrome
Keywords: leads; pacemaker; efficacy; safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Siello pacemaker lead (Experimental): Patients with Siello Pacemaker lead
  Interventions: Device: Pacemaker therapy

INTERVENTIONS:
Device: Pacemaker therapy — Implantation of the SIELLO pacemaker leads

SUMMARY:
The objective of this study is to prove the safety and efficacy of the SIELLO pacemaker leads.

DETAILED DESCRIPTION:
The assessment of the safety of SIELLO pacemaker leads is based on the collection of complications which are related to the leads. The assessment of efficacy of the SIELLO pacemaker leads is based on the collection of standard electrical lead data during the implant and follow-up procedures. Subsequent to the implantation of the SIELLO leads,five follow-up visits have been scheduled: at pre-discharge and after 1, 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Meet the indications for pacemaker therapy
* Understand the nature of the procedure
* Give informed consent
* Able to complete all testing required by the clinical protocol
* Available for follow-up visits on a regular basis at the investigational site

Exclusion Criteria:

* Meet none of the pacemaker indications
* Meet one or more of the contraindications
* Have a life expectancy of less than six months
* Cardiac surgery in the next six months -Enrolled in another cardiac clinical investigation- Have other medical devices that may interact with the implanted pacemaker

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2009-07; Primary Completion 2009-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Complication free rate of all SIELLO leads | 3 month follow-up visits
Ventricular threshold of SIELLO T (passive fixation) | 3 month follow-up visits
Atrial threshold of SIELLO S (active fixation) | 3 month follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Anselm Schaumann, Dr., Principal Investigator — n.k.
Locations (1):
- Allgemeines Krankenhaus Hamburg Altona, Hamburg, Germany